CLINICAL TRIAL: NCT06249997
Title: An Open-Label, Non-Randomized Study to Assess the Safety and Efficacy of Leniolisib in Japanese Patients With Activated Phosphoinositide 3-Kinase Delta Syndrome (APDS) Followed By An Open-Label Long-Term Extension
Brief Title: An Open-Label Study to Assess the Safety & Efficacy of Leniolisib in Japanese Patients With APDS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pharming Technologies B.V. (Industry)
Collaborators: Laboratory Corporation of America (Industry); Axial Biotech, Inc (Industry); CMIC Co, Ltd. Japan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LE 4301
Record Dates: First submitted 2023-11-21; First posted 2024-02-08 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-01

CONDITIONS: APDS Gene Mutation
MeSH Terms: interventions — leniolisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Leniolisib (Experimental): Leniolisib - Film coated tablets
  Leniolisib tablets in doses ranging from 40 to 70 mg twice daily (BID) based on body weight.
  A Part 1 clinical study report will be generated once the last patient completes the Day 85 Visit for Part 1. Patients who complete the Day 85 Visit will enter the Extension Period of the study (Part 2), in which patients will be administered leniolisib doses ranging from 40 to 70 mg BID (based on body weight) for 1 year or until marketing approval in Japan, whichever is longer. A 4-week Follow-up Period will occur after the last dose of study treatment is received.
  Interventions: Drug: Leniolisib

INTERVENTIONS:
Drug: Leniolisib — The doses selected range from 40 to 70 mg BID (based on body weight, resulting in total daily doses ranging from 80 to 140 mg a day for 12 weeks in Part I and 1 year in Part II, or until marketing approval in Japan, whichever is longer.

SUMMARY:
An Open-Label, Non-Randomized Study to Assess the Safety and Efficacy of Leniolisib in Japanese Patients With Activated Phosphoinositide 3-Kinase Delta Syndrome (APDS) Followed By an Open-Label Long-Term Extension.

For the treatment of activated phosphoinositide 3-kinase delta (PI3Kδ) syndrome (APDS).

DETAILED DESCRIPTION:
This is a 2-part, open-label, non-randomized study to assess the safety and efficacy of leniolisib in Japanese patients with APDS. At least3 patients, aged 12 to 75 years (inclusive), will be enrolled. Patient eligibility will be assessed during a 7-week Screening Period (Day -50 to Day -1). This will be followed by a 12-week Treatment Period (Part 1), in which patients will be administered leniolisib doses ranging from 40 to 70 mg twice daily (BID) based on body weight (see dose regimen table below). A Part 1 clinical study report will be generated once the last patient completes the Day 85 Visit for Part 1. Patients who complete the Day 85 Visit will enter the Extension Period of the study (Part 2), in which patients will be administered leniolisib doses ranging from 40 to 70 mg BID (based on body weight) for 1 year or until marketing approval in Japan, whichever is longer. A 4-week Follow-up Period will occur after the last dose of study treatment is received.

It is anticipated that a total of 3 patients will be enrolled into the study.

Objectives:

Part 1:

Primary:

* To assess the safety and tolerability of leniolisib
* To assess the efficacy of leniolisib on lymphoproliferation (sum of product diameters [SPD] of index lymph node lesions) and immunophenotype normalization (percentage of naïve B cells out of total B cells)

Secondary:

* To assess the efficacy of leniolisib on lymphoproliferation (non-index lymph node lesions and spleen)
* To assess the pharmacokinetics (PK) of leniolisib in the Japanese population
* To assess the efficacy of leniolisib to modify health-related quality of life
* To assess the efficacy of leniolisib by the Patient's and Physician's Global Assessments
* To assess the frequency of infections, antibiotic use, and immunoglobulin (Ig) replacement therapy and assessment of impact on other disease-related outcomes (e.g., cytopenia, colitis, and lung function)
* To assess biomarkers reflecting the efficacy of leniolisib to reduce systemic inflammatory components of the disease
* To assess the treatment benefit to individual patients

Part 2:

Primary:

- To assess the long-term safety and tolerability of leniolisib

Secondary:

* To assess the long-term efficacy of leniolisib to modify health-related quality of life
* To assess the long-term efficacy of leniolisib on lymphoproliferation (non-index lymph node lesions and spleen)

ELIGIBILITY:
Inclusion Criteria:

* Patient is Japanese.
* Patient is male or female and 12 to 75 years of age (inclusive) at the time of the first study procedure.
* Patient weighs ≥35 kg at baseline.
* Patient has a PI3Kδ genetic mutation of either the PIK3CD (APDS1) or PIK3R1 (APDS2) gene.
* Patient has at least 1 measurable nodal lesion on computed tomography (CT) or magnetic resonance imaging (MRI) scan within 6 months of Screening.
* Patient has nodal and/or extranodal lymphoproliferation and clinical findings and manifestations consistent with APDS (e.g., a history of repeated oto-sino-pulmonary infections and/or organ dysfunction consistent with APDS).
* At Screening, patient has sitting vital signs (with patient rested for at least 3 minutes) within the following ranges:
* Systolic blood pressure, 90-160 mm Hg
* Diastolic blood pressure, 50-95 mm Hg
* Pulse rate, 40-100 bpm; up to 110 bpm in adolescents

Exclusion Criteria:

- Patient has previous or concurrent use of immunosuppressive medication such as the following:

1. A mammalian target of rapamycin inhibitor (e.g., sirolimus, rapamycin, or everolimus) or a PI3Kδ inhibitor (selective or non-selective phosphoinositide 3-kinase inhibitors) within 6 weeks prior to first dose.

   - Short-term use for up to a total of 5 days is allowed but only up to 1 month prior to enrollment in the study.
2. B-cell depleters (e.g., rituximab) within 6 months prior to first dose of study treatment.

   - If patient has received prior treatment with a B-cell depleter, absolute B lymphocyte counts in the blood must have regained normal values.
3. Belimumab or cyclophosphamide within 6 months prior to first dose of study treatment.
4. Cyclosporine A, mycophenolate, 6-mercaptopurine, azathioprine, or methotrexate within 3 months prior to first dose of study treatment.
5. Glucocorticoids above 25 mg prednisone or equivalent per day within 2 weeks prior to first dose of study treatment.
6. Other immunosuppressive medications where effects are expected to persist at start of dosing of study treatment.

   * Patient has had a hematopoietic stem-cell transplant, hematopoietic cell transplant, or bone marrow transplant.
   * Patient is currently using a medication known to be a strong inhibitor or moderate or strong inducer of isoenzyme cytochrome P450 (CYP)3A if treatment cannot be discontinued or switched to a different medication prior to starting study treatment.
   * Patient is currently using medications that are metabolized by isoenzyme CYP1A2 and have a narrow therapeutic index (drugs whose exposure response indicates that increases in their exposure levels by the concomitant use of potent inhibitors may lead to serious safety concerns [e.g., Torsades de Pointes]).
   * Patient had been administered a live vaccine (this includes any attenuated live vaccines) starting from 6 weeks before the anticipated first dose of study treatment, during the treatment period, and up to 7 days after the last dose of leniolisib.
   * Patient is a pregnant or nursing (lactating) woman, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human chorionic gonadotropin laboratory test.
   * Patient is a woman of child-bearing potential, defined as a woman physiologically capable of becoming pregnant, unless she is using highly effective methods of contraception during dosing of study treatment and for 30 days after the last study procedure.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2023-08-03 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Part I: Incidence of treatment-emergent adverse events ((AEs), serious adverse events (SAEs), and AEs | Between baseline until Day 85
  Incidence of treatment-emergent adverse events (AEs), serious adverse events (SAEs), and AEs leading to discontinuation of study treatment
Part II: Long-term Incidence of treatment-emergent adverse events ((AEs), serious adverse events (SAEs), and AEs | At Day 252, through study completion, an average of 1 year
  Long-term Incidence of treatment-emergent adverse events ((AEs), serious adverse events (SAEs), and AEs leading to discontinuation of study treatment
Part I: Change from baseline in clinical laboratory test results | Between baseline until Day 85
  Number of participants with change in clinical laboratory test results (hematology, blood chemistry, urinalysis). Absolute values and change from baseline values of vital signs (including body weight) and ECG results at each visit will be listed for each patient and may be summarized using descriptive statistics. Tanner staging will be listed for each patient at each visit. Plots may also be used to display the patient data over time.
Part II: Long-term change from baseline in clinical laboratory test results | At Day 252, through study completion, an average of 1 year
  Number of participants with long-term change in clinical laboratory test results (hematology, blood chemistry, urinalysis). Absolute values and change from baseline values of vital signs (including body weight) and ECG results at each visit will be listed for each patient and may be summarized using descriptive statistics. Tanner staging will be listed for each patient at each visit. Plots may also be used to display the patient data over time.
Part I: Change from baseline in vital signs | Between baseline until Day 85
  Number of Participants with change in vital signs
Part II: Long-term change from baseline in vital signs | At Day 252, through study completion, an average of 1 year
  Number of Participants with long-term change in vital signs
Part I: Change from baseline in physical examination findings | Between baseline until Day 85
  Number of participants with change in physical examination findings
Part II: Long-term change from baseline in physical examination findings | At Day 252, through study completion, an average of 1 year
  Number of participants with long-term change in physical examination findings
Part I: Change from baseline in electrocardiograms (ECGs) | Between baseline until Day 85
  Number of participants with change in electrocardiograms (ECGs)
Part II: Long-term change from baseline in electrocardiograms (ECGs) | At Day 252, through study completion, an average of 1 year
  Number of participants with long-term change in electrocardiograms (ECGs)
Part I: To assess the efficacy of leniolisib on lymphoproliferation (SPD of index lymph node lesions) and immunophenotype normalization (percentage of naïve B cells out of total B cells) | Between baseline until Day 85
  Number of patients with change in SPD of index lesions (selected as per the Cheson methodology from magnetic resonance imaging [MRI] or computed tomography [CT] imaging) at the end of treatment
Part I: Change from baseline in the percentage of naïve B cells out of total B cells at the end of treatment | Between baseline until Day 85
  Number of participants with change in percentage of naïve B cells out of total B cells at the end of treatment

SECONDARY OUTCOMES:
Part I: Change from baseline in lymphoproliferation measured using MRI, CT imaging, or ultrasound | Between baseline until Day 85
  Parameters for change from baseline in lymphoproliferation as a secondary endpoint may include 3-dimensional (3D) volume of index and measurable non-index lesions (selected as per the Cheson methodology) and 3D volume and bi-dimensional sizes of spleen and liver, where appropriate.
Part II: Long-term change from baseline in lymphoproliferation measured using MRI, CT imaging, or ultrasound | At Day 252, through study completion, an average of 1 year
  Number of participants with change from in lymphoproliferation measured using MRI, CT imaging, or ultrasound (e.g., 3D volume of index and measurable non-index lesions [selected as per the Cheson methodology] and 3D volume and bi-dimensional sizes of spleen and liver, where appropriate) at the end of treatment.
Part I: To assess the PK of leniolisib in the Japanese population | Between baseline until Day 85
  Number of participants with change in PK parameters (including but not limited to area under the plasma concentration-time curve from time zero to 12 hours after dosing at steady state [AUC0-12,ss] and maximum plasma concentration following drug administration at steady state [Cmax,ss])
Part I: To assess the efficacy of leniolisib to modify health-related quality of life | Between baseline until Day 85
  Number of participants with change in Short Form-36 (SF-36) Survey and Work Productivity and Activity Impairment-Classroom Impairment Questionnaire (WPAI-CIQ) summary scores
Part II: To assess the long-term efficacy of leniolisib to modify health-related quality of life | At Day 252, through study completion, an average of 1 year
  Number of participants with long-term change in Short Form-36 (SF-36) Survey and Work Productivity and Activity Impairment-Classroom Impairment Questionnaire (WPAI-CIQ) summary scores
Part I: To assess the efficacy of leniolisib by the Patient's and Physician's Global Assessments | Between baseline until Day 85
  Number of participants with long-term change in visual analog scales (VAS) for Patient's and Physician's Global Assessments, measured by scale with no and maximal activity score
Part I: To assess the frequency of infections and assessment of impact on other disease-related outcomes (e.g., cytopenia, colitis, and lung function) | Between baseline until Day 85
  Number of participants with change in frequency of infections, use of antibiotics, Ig replacement therapy, and other disease complications
Part I: To assess biomarkers reflecting the efficacy of leniolisib to reduce systemic inflammatory components of the disease | Between baseline until Day 85
  Number of participants with change in High-sensitivity C-reactive protein (hsCRP), lactate dehydrogenase (LDH), beta2 microglobulin, ferritin, fibrinogen, and erythrocyte sedimentation rate
Part I: To assess the treatment benefit to individual patients | Between baseline until Day 85
  Number of patients that benefit from the treatment via narratives by the Investigator

CONTACTS AND LOCATIONS:
Overall Officials: Hirokazu Kanegane, Prof., Principal Investigator — Tokyo Medical And Dental University Hospital
Locations (2):
- Japan (2):
  - Tokyo Medical And Dental University Hospital, Tokyo, Bunkyo-ku
  - Hiroshima University Hospital, Hiroshima, Hiroshima City